CLINICAL TRIAL: NCT03959358
Title: Desensitization of Immunomodulating Agent-Related Hypersensitivity Reactions as a Means to Provide Therapeutic Options in the Management of Plasma Cell Disorders (DeHyperPCD)
Brief Title: A Study to Desensitize Allergic Reactions to Treatments for Blood Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DeHyperPCD; RV-CL-MM-PI-13170 (Other: Princess Margaret Cancer Centre)
Record Dates: First submitted 2019-05-08; First posted 2019-05-22 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Multiple Myeloma; Amyloidosis
MeSH Terms: conditions — Multiple Myeloma; Amyloidosis | interventions — Lenalidomide; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lenalidomide (Experimental): Participants will only receive lenalidomide if they had previously received this drug as a part of their treatment for multiple myeloma or amyloidosis and had experienced an allergic reaction to the drug.
  Participants will first be given a low dose of lenalidomide with increasing doses over 10-12 steps over 3.5 to 5 hours. Participants will be monitored for side effects or reactions prior to each dose step and any reactions will be managed before giving the increased dose at the next step.
  The final dose will be determined by the study doctor and is expected to be the dose that participants will restart treatment with lenalidomide at.
  Interventions: Drug: Lenalidomide
- Pomalidomide (Experimental): Participants will only receive pomalidomide if they had previously received this drug as a part of their treatment for multiple myeloma or amyloidosis and had experienced an allergic reaction to the drug.
  Participants will first be given a low dose of pomalidomide with increasing doses over 10-12 steps over 3.5 to 5 hours. Participants will be monitored for side effects or reactions prior to each dose step and any reactions will be managed before giving the increased dose at the next step.
  The final dose will be determined by the study doctor and is expected to be the dose that participants will restart treatment with pomalidomide at.
  Interventions: Drug: Pomalidomide

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide is an antineoplastic and immunomodulatory agent that will be given as a liquid in syringes to be taken orally (by mouth).
  Other Names: REVLIMID
  Arms: Lenalidomide
Drug: Pomalidomide — Pomalidomide is an antineoplastic and immunomodulatory agent that will be given as a liquid in syringes to be taken orally (by mouth).
  Other Names: POMALYST
  Arms: Pomalidomide

SUMMARY:
Patients with multiple myeloma (a type of blood cancer affecting the white blood cells) or amyloidosis (abnormal buildup of a protein called amyloid in the body) are often given treatment with the drugs lenalidomide or pomalidomide. Some patients may experience an allergic reaction to these drugs which would mean stopping the treatment.

The purpose of this research study is to see how safe and useful desensitization is in allowing patients to receive further treatment with lenalidomide or pomalidomide.

DETAILED DESCRIPTION:
Some doctors believe that the body may be taught to react less or stop reacting to, the things that would otherwise trigger an allergic reaction. This is called desensitization. Desensitization is usually done with repeat exposure to the thing that causes the allergic reaction. For example, people who have allergies may receive small, controlled doses of the allergen over a period of time until the allergic reactions are tolerable or are stopped completely.

The researchers want to see if giving low doses of lenalidomide or pomalidomide to people who experienced an allergic reaction to these medications can become desensitized so that they are able to continue treatment for their disease with these drugs.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Adult patients 18 years old or older
* All study participants must be registered into the mandatory Lenalidomide or Pomalidomide Pregnancy Prevention Plan, and be willing and able to comply with the requirements.
* Females of reproductive potential must adhere to the pregnancy testing and contraceptive techniques as required by the Pregnancy Prevention Plan.
* Patient diagnosed with multiple myeloma or amyloidosis, with history of HSR to lenalidomide or pomalidomide, who had experienced moderate-severe (Grade ≥2 CTCAE v5.0) cutaneous reactions to IMiDs, with or without being symptomatic (itchy rash). Patients who developed HSR to IMiDs (lenalidomide or pomalidomide) will be assessed according to the CTCAE v 5.0 grading criteria during enrolment, and the severity of the grading (Grade ≥ 2 or otherwise) is recorded for the purpose of future subgroup analysis. OR
* Complained of angioedema or anaphylaxis reactions attributable to lenalidomide or pomalidomide.
* Patients must be afebrile at least 48 hours prior to proposed desensitization day.
* For patients with existing body rash, a complete resolution of rash is needed prior to Rapid Desensitization Program procedures at least 7 days prior to desensitization.
* Patients may continue to administer their current medication prior to the start of Rapid Desensitization Program (RDP). Best possible medication history will be taken prior to RDP, with the exception of withholding beta- blockers on the day of desensitization. Patient's allergy history will be documented.

Exclusion Criteria:

* Female who is pregnant or suspected of being pregnant or breast feeding or likely to breast feed during the study duration
* Inability to take oral medications.
* History of Steven-Johnson Syndrome (SJS), Toxic Epidermal Necrolysis (TEN) and Drug Reaction with Eosinophilia and Systemic Symptoms (DRESS).
* Patients who are taking IMiDs-based therapy for an indication other than multiple myeloma (MM) and/or systemic amyloidosis (AL).
* The development of erythema nodosum, if characterized by a desquamating rash while taking thalidomide, IMiDs or similar drugs.
* Active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B virus vaccine or previous infection (HepB core Ab +, but HepB sAg negative) are eligible.
* Patients who, for whatever reason, are unable to tolerate IMiDs (other than hypersensitivity reactions).
* Patients who have completed 3 RDPs and continued to have breakthrough hypersensitivity reactions (HSR) post Rapid Desensitization Program (RDP).
* Patients who had experienced IMiDs-related hypersensitivity reaction that is less than Grade 2 (Grade 1) as per CTCAE v5.0.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Number of participants successfully completing desensitization program | 12 days

SECONDARY OUTCOMES:
Distress Assessment and Response Tool (DART) score | 90 days post desensitization program
  Rating of physical symptoms, practical concerns, and emotional concerns on a scale from 1-10. 0 = no symptoms/concerns, 10=worse possible experience of the symptom/concern
Edmonton Symptom Assessment System (ESAS) score | 90 days post desensitization program
  A rating of nine common symptoms on a scale from 0-10. 0 = no symptoms, 10=worse possible experience of the symptom
Frequency of interrupted treatment with immunomodulating agent | 90 days post desensitization program
Duration of interrupted treatment with immunomodulating agent | 90 days post desensitization program
Mortality rate associated with disease progression or treatment-related toxicity | 90 days post desensitization program
Frequency of rash recurrence | 90 days post desensitization
Duration of treatment with immunomodulating agent post desensitization | 90 days post desensitization
Incidence of adverse events during desensitization procedures and hospital stay | 12 days
Total duration of treatment with immunomodulating agent | 90 days post desensitization
Duration of treatment with supportive care agents | 90 days post desensitization

CONTACTS AND LOCATIONS:
Overall Officials: Anca Prica, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada